CLINICAL TRIAL: NCT04820985
Title: Analyse de la Composition du Microbiote Vaginal à différents Temps de la Prise en Charge en FIV et corrélation Avec le Taux de progestérone sérique le Jour du Transfert d'Embryon
Brief Title: Analysis of the Composition of the Vaginal Microbiota During IVF Treatment and Correlation With Serum Progesterone Level on the Day of Embryo Transfer
Acronym: MICROFIV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2020-01/SH-01
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: IVF
Keywords: Pregnancy; vaginal microbiota; Progesterone
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women undergoing IVF
  Interventions: Other: Vaginal swab; Other: Blood test

INTERVENTIONS:
Other: Vaginal swab — Vaginal flora swab 3 months before stimulation, at oocyte puncture, embryo transfer and beta-human chorionic gonadotropin dosing
Other: Blood test — Blood sample to measure plasma dose of progesterone

SUMMARY:
The composition of the vaginal microbiota varies throughout a woman's life and is sensitive to hormonal and environmental factors. Specifically, hormonal treatments necessary in the medically assisted procreation (MAP) processes can influence the vaginal microbiota. New sequencing techniques have been used to characterize the vaginal microbiota, demonstrating that the microbiota could be divided into 5 classes. The composition of the vaginal microbiota seems to have an implication in the evolution of a pregnancy after IVF. It is therefore essential to have more data on the evolution of the vaginal microbiota at the different stages of IVF treatment and to analyze whether this evolution can be predictive of the success of embryo implantation. Good endometrial progesterone impregnation is an essential prerequisite for ensuring embryo implantation. Indeed, supporting the luteal phase through vaginal progesterone is an essential step in IVF protocols to ensure synchronization between endometrial maturation and embryonic age. However, the serum progesterone level on the day of embryo transfer varies widely between patients. Several factors such as age, vaginal mucosa trophicity, estrogen impregnation and sexual activity are known to affect the vaginal absorption of progesterone. The treatments and vaginal examinations performed during the IVF procedure could also have an impact on the constitution of the vaginal microbiota. The hypothesis of this research is that there is an alteration in the vaginal microbiota during the IVF process which may alter the absorption of vaginal progesterone, with an impact on the failure or success of embryo implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient in round 1 or 2 of IVF or IVF-ICSI with transfer of a fresh embryo with a normal preimplantation assessment, without antibiotic treatment in the 3 months preceding the sample.
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* Use of antibiotics in the 3 months preceding the sample.
* Patient presenting an anomaly in the implantation assessment.
* Presence of uterine malformation, hydrosalpinx, chronic vaginosis.
* Patient undergoing a protocol to study endometrial receptivity.
* Patient of African American, African or Latin American origin (patients born to two parents of Hispanic origin) as people of African and Hispanic origin have a type IV flora vs people of Caucasian origins who have type I, II, III and V of the Ravel classification .
* Cancellation of the procedure for various reasons (stimulation failure, collection failure, fertilization failure or embryonic segmentation).
* Patient taking a freeze-all approach (freezing of the embryos) for various causes (risk of ovarian hyperstimulation, increase in progesterone, too thin endometrium, etc.).
* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Patients aged 18 to 40 inclusive, Round1 or 2 of IVF or IVF-ICSI with fresh embryo transfer, without taking antibiotics in the 3 months preceding the first sample treated in the AMP center of the CHU de Nîmes.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Class of vaginal flora according to community state type | 3 Months before ovarian stimulation
  Classified into 5 classes of vaginal flora described according to Smith & Ravel 2017
Microbiota richness of vaginal flora | 3 Months before ovarian stimulation
  Measured by operational taxonomic unit
Microbiota alpha diversity of vaginal flora | 3 Months before ovarian stimulation
  Shannon Index
Microbiota beta diversity of vaginal flora | 3 Months before ovarian stimulation
  Bray Curtis index
Plasma progesterone level on the day of embryo transfer | Day of embryo transfer (Day 0)
  Measured by chemiluminescence (nmol/L)

SECONDARY OUTCOMES:
Class of vaginal flora according to community state type | Day of oocyte puncture (Month 3)
  Classified into 5 classes of vaginal flora described according to Smith & Ravel 2017
Class of vaginal flora according to community state type | Day of embryo transfer (Day 93)
  Classified into 5 classes of vaginal flora described according to Smith & Ravel 2017
Class of vaginal flora according to community state type | Day of beta-human chorionic gonadotropin dosage (Day 108)
  Classified into 5 classes of vaginal flora described according to Smith & Ravel 2017
Microbiota richness of vaginal flora | Day of oocyte puncture (Month 3)
  Measured by operational taxonomic unit
Microbiota richness of vaginal flora | Day of embryo transfer (Day 93)
  Measured by operational taxonomic unit
Microbiota richness of vaginal flora | Day of beta-human chorionic gonadotropin dosage (Day 108)
  Measured by operational taxonomic unit
Microbiota alpha diversity of vaginal flora | Day of oocyte puncture (Month 3)
  Shannon Index
Microbiota alpha diversity of vaginal flora | Day of embryo transfer (Day 93)
  Shannon Index
Microbiota alpha diversity of vaginal flora | Day of beta-human chorionic gonadotropin dosage (Day 108)
  Shannon Index
Microbiota beta diversity of vaginal flora | Day of oocyte puncture (Month 3)
  Bray Curtis index
Microbiota beta diversity of vaginal flora | Day of embryo transfer (Day 93)
  Bray Curtis index
Microbiota beta diversity of vaginal flora | Day of beta-human chorionic gonadotropin dosage (Day 108)
  Bray Curtis index
Pregnancy success | Month 3
  Yes/No
Pregnancy progression | Month 3
  Implantation failure/progression/miscarriage
Treatments received for IVF | Month 3
  Description of treatments, taken from patient file
Plasma progesterone level | Month 3
  Measured by chemiluminescence (nmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Huberlant, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nimes, Nîmes, France

REFERENCES:
- [Background] Smith SB, Ravel J. The vaginal microbiota, host defence and reproductive physiology. J Physiol. 2017 Jan 15;595(2):451-463. doi: 10.1113/JP271694. Epub 2016 May 5. PMID 27373840